CLINICAL TRIAL: NCT00545116
Title: Short-term Effects of Hesperidin on Bone Biomarkers in Postmenopausal Women: a Randomized Placebo-controlled Trial
Brief Title: Effects of Hesperidin on Bone Biomarkers in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nestec 06.34
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2014-01

CONDITIONS: Osteopenia; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- a (Experimental): Active carrier 1: biscuit providing 250 mg hesperidin per piece(6g)
  Interventions: Other: Hesperidin
- b (Experimental): Active carrier 2: liquid skim milk providing 250 mg hesperidin/serve (200 ml) and containing around 300 mg calcium/serving
  Interventions: Other: Hesperidin
- c (Placebo Comparator): Placebo carrier 1: biscuit with the same nutrient composition and appearance as the active biscuit carrier but minus hesperidin
  Interventions: Other: Hesperidin
- d (Placebo Comparator): Placebo carrier 2: liquid skim milk with the same nutrient composition and appearance as the active milk carrier but minus hesperidin
  Interventions: Other: Hesperidin

INTERVENTIONS:
Other: Hesperidin — 250 mg of hesperidin twice a day taken oraly in a biscuit or in milk for 6 months

SUMMARY:
The primary objective of this clinical trial is to determine the effects of hesperidin on biochemical markers of bone in post-menopausal women.

The secondary objectives are:

* To investigate changes in bone formation and bone resorption markers in response to hesperidin intake
* To compare the efficacy of hesperidin in a milk versus biscuit
* To collect safety information of hesperidin consumption in a human trial

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling women
* More than 4 years post-menopause (natural or surgical)
* Generally healthy as determined by standard medical assessment on physical and mental health
* Willing to comply with the study procedures
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data
* Having received both oral and written explanations about the study
* Having provided her written informed consent

Exclusion Criteria:

* Intestinal or severe metabolic diseases / disorders such as diabetes, renal, hepatic or pancreatic diseases / disorders, ulcer, hyperthyroidism, malignance, chronic malnutrition
* Have had major gastrointestinal surgery
* On therapy with drugs known to interfere with bone metabolism such as steroids, vitamin D or its derivatives, bisphosphonates, strontium ranelate, PTH, calcitonin, raloxifene, etc.
* Had sustained a fracture in the preceding 12 months
* On hormone replacement therapy (HRT) in the previous 3 months before entering the study
* Taking medications containing hesperidin (e.g.Daflon) or known to interfere with hesperidin (statins, therapy for circulatory disorders, anti-depressants)
* Known to have allergic reactions to citrus-containing foods
* Baseline calcium intake less than 500 mg/day
* Have an alcohol intake > 2 glasses of wine per day (3dL/day), or > 2 beers (3dL/d) or > 1 shot glass of hard alcohol
* Heavy smoker (more than 10 cigs a day)
* Special dietary habits (vegetarians)
* Phytoestrogens or antioxidants (dietary supplements) consumption

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline for bone formation (serum P1NP & osteocalcin) and bone resorption (urinary NTX & serum CTX) markers | Six months

SECONDARY OUTCOMES:
Full blood biochemistry analyses including lipid profile | 6 months
Percentage change from baseline for osteoarthritis markers (CTX2 and others) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Chee, PhD, Principal Investigator — Faculty of Allied Health Sciences, UKM
Locations (1):
- Hospital of UKM, National University of Malaysia, Kuala Lumpur, Malaysia